CLINICAL TRIAL: NCT03475069
Title: Effects of a Special Exercise Program on Physical Function and Quality of Life Versus Plates and Calisthenics Exercises on Patients With Type 2 Diabetes Mellitus
Brief Title: Which Exercises Should Diabetic Patients do?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Başar Öztürk, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: drskull78
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Type2 Diabetes; Physical Activity
Keywords: Type 2 Diabetes Mellitus; Exercise; Physical Performance; Physiological Cost Index
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual intervention (Experimental): This exercise program was prepared specific to each patient in this group according to his/her physiotherapy assessment, functional performance tests and body analysis results. This exercise type focuses on patients' physical demands. Exercises were applied by a researcher physiotherapist.
  Interventions: Other: Custom Designed Exercises
- Plates intervention (Experimental): Plates exercises were applied as a group treatment. This exercise type contains non-impact exercises to develop strength, flexibility, balance, and inner awareness.Plates exercises were applied as a group treatment. Exercises were applied by a researcher physiotherapist.
  Interventions: Other: Plates Exercises
- Chalistenics intervention (Experimental): These exercises included range of motion exercises of neck (flexion, extension, lateral flexion and rotation), shoulder (flexion, extension, abduction, adduction, internal and external rotation), elbow (flexion and extension), forearm (pronation and supination), wrist (flexion and extension), hip (flexion, extension, abduction and adduction, internal and external rotation), knee (flexion and extension), foot (dorsi and plantar flexion, pronation and supination) and trunk (flexion, extension, lateral flexion and rotation). Exercises were applied by a researcher physiotherapist.
  Interventions: Other: Calisthenics Exercises

INTERVENTIONS:
Other: Custom Designed Exercises
  Arms: Individual intervention
Other: Plates Exercises
  Arms: Plates intervention
Other: Calisthenics Exercises
  Arms: Chalistenics intervention

SUMMARY:
Type 2 Diabetes Mellitus (DM) is a widespread worldwide disease. Exercise therapy is an effective method but which exercise types are more effective is an important question.

This study was designed to compare the effects of three different exercise programs on physical function and quality of life in Type 2 DM. Forty-two patients with Type 2 DM participated in the study. The patients were randomly assigned to three groups. Client based exercises in accordance with physiotherapy assessment were applied to group 1 (aged 51.42±4.60 years; body mass index 35.28±4.21 kg/m² kg/m²), Clinical Plates exercises were applied to group 2 (aged 53.07 ±5.12 years; body mass index 35.56±4.83 kg/m²) and a standard program including calisthenics exercises were applied to group 3 for 12 weeks, 3 days a week. 6 minutes walk test (6 MWT) and physiological cost index (PCI), timed up and go test (TUG) and SF-36 quality of life questionnaire were performed before and after the 12-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can walk independently.
* Patients who accept doing exercises for 12 weeks, 3 days a week properly Patients whose cognitive status are enough for understanding and realizing different exercise types.

Exclusion Criteria:

* Patients with orthopaedic or surgical problems that prevent walking.
* Patients with neuropathy that prevent walking.
* Patients who have foot ulcers.
* Patients with neurological problems.
* Patients with cardiac, pulmonary and systematic problems that cause contraindication for exercise.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-10-20 (Actual); Primary Completion 2013-12-15 (Actual); Study Completion 2014-02-16 (Actual)

PRIMARY OUTCOMES:
Energy expenditure after physical performance | 3 months
  Physiological cost index (PCI) calculated during 6 minutes walk test (6MWT) after exercise period. PCI is a clinical tool thought to indicate the energy expenditure. Subjects walk at their preferred pace, usually following a track of known distance, while heart rate and time are noted. After measurement of resting heart rate, a person's PCI in beats per meter is calculated. 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. Mean PCI values for healthy adults have been reported to be between 0.23 and 0.42 beat/meter. The energy consumption increases as the number increases and it indicates fatigue. Lower than 0.23 indicates low energy consumption and is not considered normal.
Quality of life | 3 months
  The 36-Item Short Form Health Survey (SF-36) questionnaire was applied after exercise period. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. The test consists of 36 questions and requires 10 minutes to administer. The Sf-36 includes a multi-item scale with 8 subscales. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section.
  Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
  Sections:
  Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health.

SECONDARY OUTCOMES:
Timed up and go test | 3 months
  Standing, walking and sitting performance were measured after exercise period by timed up and go test (TUG). TUG is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. ≤10 seconds=normal, ≤ 20 seconds=good mobility, can go out alone, mobile without gait aid, ≤ 30 seconds=problems, can not go outside alone, requires gait aid.
Body mass index | 3 months
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women. It was measured by bioelectrical impedance device.
  A BMI below 18.5 is considered underweight. A BMI of 18.5 to 24.9 is considered healthy. A BMI of 25 to 29.9 is considered overweight. A BMI of 30 or higher is considered obese.

CONTACTS AND LOCATIONS:
Locations (1):
- Başar Öztürk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided